CLINICAL TRIAL: NCT01200108
Title: A Double-Blind, Randomized, Placebo-Controlled Trial to Evaluate Tolerability, Safety and Efficacy of AKITA Inhaled Steroid Suspension for Inhalation (AICS) in Subjects With Asthma Requiring Chronic Oral Corticosteroid Treatment
Brief Title: AKITA Inhaled Steroid Suspension for Inhalation (AICS) in Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Activaero GmbH (Industry)
Responsible Party: Dr. Thomas Hofmann, Activaero GmbH
Other Study IDs: Acti-AICS-001
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Asthma
Keywords: Severe Asthma, requiring chronic oral steroid use
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Budesonide high dose via AKITA (1mg/2ml) (Experimental)
  Interventions: Drug: Budesonide
- Budesonide low dose via AKITA (0.5mg/2ml) (Experimental)
  Interventions: Drug: Budesonide
- Budesonide high dose via conventional nebulizer (1mg/2ml) (Active Comparator)
  Interventions: Drug: Budesonide
- Placebo via AKITA (No Intervention)

INTERVENTIONS:
Drug: Budesonide
  Arms: Budesonide high dose via AKITA (1mg/2ml)
Drug: Budesonide
  Arms: Budesonide low dose via AKITA (0.5mg/2ml)
Drug: Budesonide
  Arms: Budesonide high dose via conventional nebulizer (1mg/2ml)

SUMMARY:
The goal of treatment with AICS is weaning from oral corticosteroids, i.e. a reduction of the oral corticosteroid dose. An anticipated treatment benefit of AICS is a reduction of oral corticosteroid dose and stability/improvement of clinical parameters related to asthma in the targeted subject population. Ultimately, the goal is to free subjects with severe asthma from the burden of chronic oral steroid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to the performance of any study-related procedures
* Age ≥ 18 and ≤ 65 year of age Diagnosis of asthma (ATS definition, either allergic or non-allergic) for ≥ 6 months
* Asthma treated for at least 3 months with inhaled (ICS) and oral corticosteroids (OCS). Exact baseline level will be measured during the screening period by subject diary entries
* FEV1 ≥ 40% or ≤ 79% predicted at the Screening or Baseline Visit
* Documented increase of FEV1 within 15-30 minutes after the use of inhaled Salbutamol at the Screening Visit or within 2 years prior to Screening
* Mandatory usage of long-acting β-agonists
* A negative pregnancy test must be available for any women of childbearing potential at screening and, in addition, a negative urine pregnancy test must be present at randomization (prior to randomization to one of the treatment groups!)
* Women of childbearing potential must agree to use a reliable method of contraception from the screening until 4 weeks after study completion or after study drug discontinuation in case study drug treatment is stopped prematurely. - In this study, hormone-based contraceptives alone are not considered as reliable method

Exclusion Criteria:

* History of allergy or adverse experience with Budesonide
* Pregnant women or nursing mothers
* Upper respiratory tract infection within 4 weeks of Screening
* Emergency room visit for treatment of asthma exacerbation within 4 weeks of Screening
* Hospitalization for asthma within 3 months of Screening
* Use of anti-IgE, methotrexate, oral gold, Dapsone, or i.v. gamma globulin within 3 months of Screening
* Treatment with other investigational asthma treatment within 30 days prior to Screening
* Evidence of chronic lung diseases other than asthma, including but not limited to: cystic fibrosis, allergic bronchopulmonary aspergillosis (ABPA), COPD, chronic bronchitis and emphysema
* History of medication noncompliance
* History of significant medical illness or condition that in the Investigator's opinion places the subject at undue risk by participating in the study
* Past episode of anaphylaxis with severe respiratory symptoms
* Oral corticosteroid average daily dose exceeding a maximum amount
* Currently smoking or history of smoking ≥ 10 pack years
* Taking oral or i.v. corticosteroids for any disease indication other than asthma
* Abnormal lab values for chemistry tests at Screening that may indicate impaired ability to metabolize and/or excrete Budesonide (AST, ALT > 3 times upper limit of normal range, serum creatinine > 1.5 times upper limit of normal range)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kardos, MD, Principal Investigator — Peter Kardos
Locations (23):
- Germany (9):
  - Berlin
  - Bonn
  - Darmstadt
  - Peter, Kardos, MD, Frankfurt
  - Marburg
  - München
  - Rodgau-Dudenhofen
  - Rüdersdorf
  - Schwetzingen
- Poland (8):
  - Katowice
  - Krakow
  - Lódz
  - Lublin
  - Poznán
  - Skierniewice
  - Warsaw
  - Wroclaw
- Ukraine (6):
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Vinnytsia

REFERENCES:
- See also: Homepage of the trial sponsor — http://www.activaero.de